CLINICAL TRIAL: NCT02104466
Title: Randomized Controlled Pilot Trial of Adjunct Group Acupuncture vs Usual Care Among Patients With Painful Diabetic Neuropathy
Brief Title: Group Acupuncture Treatment Effects for Painful Diabetic Neuropathy (GATE-PDN)
Acronym: GATE-PDN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-12822; K01AT006545 (NIH)
Record Dates: First submitted 2014-03-27; First posted 2014-04-04 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: acupuncture; pain; neuropathy
MeSH Terms: conditions — Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment as Usual (TAU) (No Intervention): Participants randomized to this arm will receive usual care with no acupuncture.
- TAU + 12 wks of acupuncture 1x/week (Experimental): Participants randomized to this arm will receive usual care with adjunctive acupuncture once per week for a period of 12 weeks.
  Interventions: Procedure: Acupuncture
- TAU + 12 wks of acupuncture 2x/week (Experimental): Participants randomized to this arm will receive usual care with adjunctive acupuncture twice per week for a period of 12 weeks.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture will be delivered in a group setting, in a common space with multiple reclining chairs. The initial acupuncture treatment will include a one-on-one diagnostic interview with one of the study acupuncturists for up to 30 minutes, followed by administration of acupuncture needles retained for 20-40 minutes. For subsequent group acupuncture treatments, participants will have a 10-15 minute diagnostic intake with the acupuncturist, followed by administration of acupuncture needles retained for 20-40 minutes. Eight to twelve needles will be administered in acupuncture points selected based on a treatment manual developed for the study. All treatments will be administered using sterile, disposable, surgical stainless steel acupuncture needles.
  Arms: TAU + 12 wks of acupuncture 1x/week; TAU + 12 wks of acupuncture 2x/week

SUMMARY:
Peripheral neuropathy is a common complication of diabetes, and one of the strongest determinants of reduced health-related quality of life among people with diabetes. Neuropathy frequently presents with painful symptoms, activity limitation, insomnia, fatigue, and depressive symptoms. Anti-convulsants and tricyclic anti-depressants provide at least moderate pain relief for 25-50% of patients with painful diabetic neuropathy (PDN), but often decrease other domains of quality of life through adverse effects, such as dry mouth, dizziness, nausea, drowsiness, and urinary problems. Effective, non-pharmaceutical approaches for PDN are needed, particularly for low income and racial/ethnic minorities who are at highest risk of diabetes and related complications. Acupuncture is a promising treatment for PDN, but evidence is limited. To address the significant public health need related to pain management among underserved people with diabetes, this study proposes an innovative, group-based model of acupuncture for PDN at an urban safety net hospital. Sixty patients who have PDN will be enrolled and randomized to one of three arms: (a) usual care combined with 12 weeks of group acupuncture twice weekly, (b) usual care combined with 12 weeks of group acupuncture once weekly, or (c) usual care alone (20 in each group). The aims of the study are to determine the feasibility of group acupuncture for PDN among underserved patients with diabetes; to evaluate the preliminary treatment effects of group acupuncture on pain, health-related quality of life, depressive symptoms, sleep disturbance, nerve conduction velocity, and protective sensation; and to determine the optimal frequency of acupuncture treatments.

The investigators hypothesize that compared to patients receiving usual care alone, patients who undergo weekly group acupuncture treatments will have:

1. decreased pain intensity
2. improved health-related quality of life
3. improved sural nerve conduction velocity

ELIGIBILITY:
Inclusion Criteria:

* English, Spanish, or Cantonese speaking
* Diagnosed with type 2 diabetes mellitus
* Distal lower limb pain present for at least three months
* A score of 4 or greater on the 11-point Pain Intensity Numerical Rating Scale (PI-NRS) for the pain of diabetic peripheral neuropathy at least four days a week before randomization
* Pain characterized as burning, shooting, or stabbing in nature
* Ability to understand study procedures and willingness to comply with them for the entire length of the study
* A score of less than 8 on the Semmes-Weinstein monofilament test
* Stable use of pain control medications for PDN in the one month prior to screening (e.g. no change in prescription) or no use of pain control medications for PDN within the past one month

Exclusion Criteria:

* Substance abuse (as assessed by the Simple Screening Instrument for Substance Abuse)
* Unstable medical condition (e.g. severe pulmonary disease, myocardial infarction, severe depressive symptoms)
* Electrical therapy (e.g. TENS unit) or patch treatment (e.g. lidocaine or capsaicin) for PDN used within the past two weeks
* Acupuncture, moxibustion, cupping or herbal medicine for PDN used within the past two weeks
* Pregnancy, planning a pregnancy or breast-feeding
* Inability or unwillingness to comply with this study protocol, assessed prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percentage of recruited participants retained for the 12-week intervention period | 12 weeks
Change from baseline in average weekly pain on the 11-point Pain Intensity Numerical Rating Scale (PI-NRS) at week 12 | Baseline, Weeks 1-12

SECONDARY OUTCOMES:
Pain Qualities Assessment Scale | Baseline, Weeks 1-12, Week 24
Health-related quality of life | Baseline, Week 6, Week 12, Week 18
  The following questionnaires will be used: Norfolk Quality of Life Questionnaire - Diabetic Neuropathy; Diabetes Distress Scale; Brief Pain Inventory Interference Scale; Centers for Disease Control and Prevention Healthy Days Measure
Depressive symptoms using the Patient Health Questionnaire | Baseline, Week 6, Week 12, Week 18
Participant rating of global improvement using the Patient Global Impression of Change scale | Week 12
Patient-centered symptom severity using the Measure Yourself Medical Outcome Profile | Baseline, Week 6, Week 12, Week 18
NIH PROMIS Sleep Disturbance Scale | Baseline, Week 6, Week 12, Week 18
Protective sensation of the feet using a 5.07 Semmes-Weinstein monofilament | Baseline, Week 12, Week 18
Patient satisfaction | Week 12
  At Week 12, an exit interview will be administered to inquire about satisfaction with the acupuncture services and study procedures.

OTHER OUTCOMES:
Use of medications at baseline and throughout 12-week intervention period | Baseline, Week 12
  Data about medication use will be extracted from the participant's medical chart, including type(s) of analgesics, total dose, and the number of agents.

CONTACTS AND LOCATIONS:
Overall Officials: Maria T Chao, DrPH, MPA, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Solli O, Stavem K, Kristiansen IS. Health-related quality of life in diabetes: The associations of complications with EQ-5D scores. Health Qual Life Outcomes. 2010 Feb 4;8:18. doi: 10.1186/1477-7525-8-18. PMID 20132542
- [Background] Van Acker K, Bouhassira D, De Bacquer D, Weiss S, Matthys K, Raemen H, Mathieu C, Colin IM. Prevalence and impact on quality of life of peripheral neuropathy with or without neuropathic pain in type 1 and type 2 diabetic patients attending hospital outpatients clinics. Diabetes Metab. 2009 Jun;35(3):206-13. doi: 10.1016/j.diabet.2008.11.004. Epub 2009 Mar 17. PMID 19297223
- [Background] Jensen MP, Chodroff MJ, Dworkin RH. The impact of neuropathic pain on health-related quality of life: review and implications. Neurology. 2007 Apr 10;68(15):1178-82. doi: 10.1212/01.wnl.0000259085.61898.9e. PMID 17420400
- [Background] Vinik A. CLINICAL REVIEW: Use of antiepileptic drugs in the treatment of chronic painful diabetic neuropathy. J Clin Endocrinol Metab. 2005 Aug;90(8):4936-45. doi: 10.1210/jc.2004-2376. Epub 2005 May 17. PMID 15899953
- [Background] Wong MC, Chung JW, Wong TK. Effects of treatments for symptoms of painful diabetic neuropathy: systematic review. BMJ. 2007 Jul 14;335(7610):87. doi: 10.1136/bmj.39213.565972.AE. Epub 2007 Jun 11. PMID 17562735
- [Background] Wiffen P, Collins S, McQuay H, Carroll D, Jadad A, Moore A. Anticonvulsant drugs for acute and chronic pain. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD001133. doi: 10.1002/14651858.CD001133.pub2. PMID 16034857
- [Background] Saarto T, Wiffen PJ. Antidepressants for neuropathic pain. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD005454. doi: 10.1002/14651858.CD005454.pub2. PMID 17943857
- [Background] Rutkove SB. A 52-year-old woman with disabling peripheral neuropathy: review of diabetic polyneuropathy. JAMA. 2009 Oct 7;302(13):1451-8. doi: 10.1001/jama.2009.1377. Epub 2009 Sep 8. PMID 19738078
- [Background] Adams AS, Zhang F, Mah C, Grant RW, Kleinman K, Meigs JB, Ross-Degnan D. Race differences in long-term diabetes management in an HMO. Diabetes Care. 2005 Dec;28(12):2844-9. doi: 10.2337/diacare.28.12.2844. PMID 16306543
- [Background] Karter AJ, Ferrara A, Liu JY, Moffet HH, Ackerson LM, Selby JV. Ethnic disparities in diabetic complications in an insured population. JAMA. 2002 May 15;287(19):2519-27. doi: 10.1001/jama.287.19.2519. PMID 12020332
- [Derived] Chao MT, Schillinger D, Nguyen U, Santana T, Liu R, Gregorich S, Hecht FM. A Randomized Clinical Trial of Group Acupuncture for Painful Diabetic Neuropathy Among Diverse Safety Net Patients. Pain Med. 2019 Nov 1;20(11):2292-2302. doi: 10.1093/pm/pnz117. PMID 31127837